CLINICAL TRIAL: NCT03257644
Title: An Open-Label, Pilot Pharmacokinetic Study of Ruxolitinib Phosphate Cream in Pediatric Subjects With Atopic Dermatitis
Brief Title: A Pharmacokinetic Study of Ruxolitinib Phosphate Cream in Pediatric Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-102
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Janus kinase (JAK) inhibitor; pediatric; inflammation
MeSH Terms: conditions — Dermatitis, Atopic; Inflammation | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): Ruxolitinib phosphate cream 0.5%.
  Interventions: Drug: Ruxolitinib phosphate cream
- Cohort 2 (Experimental): Ruxolitinib phosphate cream 1.5%.
  Interventions: Drug: Ruxolitinib phosphate cream
- Cohort 3 (Experimental): Ruxolitinib phosphate cream 0.75%.
  Interventions: Drug: Ruxolitinib phosphate cream
- Cohort 4 (Experimental): Ruxolitinib phosphate cream 1.5%.
  Interventions: Drug: Ruxolitinib phosphate cream
- Cohort 5 (Experimental): Ruxolitinib phosphate cream 0.75%.
  Interventions: Drug: Ruxolitinib phosphate cream
- Cohort 6 (Experimental): Ruxolitinib phosphate cream 1.5%.
  Interventions: Drug: Ruxolitinib phosphate cream

INTERVENTIONS:
Drug: Ruxolitinib phosphate cream — Ruxolitinib phosphate cream at the protocol-defined dose strength based on cohort assignment.
  Other Names: INCB018424

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and the pharmacokinetics (PK) of topical ruxolitinib cream applied to pediatric subjects (age ≥ 2 to 17 years) with atopic dermatitis (AD).

DETAILED DESCRIPTION:
Study has been modified to include younger pediatric subjects (age ≥2 to 11) in four additional cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects aged ≥ 2 to 17 years, inclusive
* Subjects diagnosed with AD as defined by the Hanifin and Rajka criteria.
* Subjects with active inflammation associated with AD.
* Subjects with an Investigator's Global Assessment (IGA) score of at least 2 at screening and baseline.
* Subjects with body surface area (BSA) of AD involvement of 8% to 20% at screening and baseline.
* Subjects who agree to discontinue all agents used to treat AD from screening through the final follow-up visit.
* Subjects of childbearing potential must agree to take appropriate precautions to avoid pregnancy or fathering a child for the duration of study participation.
* Written informed consent of the parent(s) or legal guardian and a verbal or written assent from the subject when possible.

Exclusion Criteria:

* Unstable course of AD (spontaneously improving or rapidly deteriorating) as determined by the investigator over the previous 4 weeks before baseline.
* Use of topical treatments for AD (other than bland moisturizer such as Eucerin® cream) within 2 weeks of baseline.
* Concurrent conditions and history of other diseases:

  * Presence of AD lesions only on the hands or feet without a history of involvement of other classical areas of involvement such as the face or the flexural folds.
  * Other types of eczema.
  * Any other concomitant skin disorder (eg, generalized erythroderma such as Netherton Syndrome, or psoriasis), pigmentation, or extensive scarring that in the opinion of the investigator may interfere with the evaluation of AD lesions or compromise subject safety.
  * Immunocompromised (eg, lymphoma, acquired immunodeficiency syndrome, Wiskott-Aldrich syndrome) or have a history of malignant disease within 5 years before the baseline visit.
  * Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks before the baseline visit.
  * Active acute bacterial, fungal, or viral (eg, herpes simplex, herpes zoster, chicken pox) skin infection within 1 week before the baseline visit.
  * Chronic asthma requiring more than 880 μg of inhaled budesonide or equivalent high dose of other inhaled corticosteroids.
* Subjects with cytopenias at screening per protocol-defined criteria.
* Use of the following medications:

  * Systemic immunosuppressive or immunomodulating drugs (eg, oral or injectable corticosteroids, methotrexate, cyclosporine, mycophenolate mofetil, azathioprine) within 4 weeks or 5 half-lives of baseline (whichever is longer).
  * Subjects taking potent systemic cytochrome P450 3A4 inhibitors or fluconazole within 2 weeks or 5 half lives, whichever is longer, before the baseline visit (topical agents with limited systemic availability are permitted).
  * Subjects who have previously received JAK inhibitors, systemic or topical (eg, ruxolitinib, tofacitinib, baricitinib, filgotinib, lestaurtinib, pacritinib).
  * Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before the baseline visit with another investigational medication or current enrollment in another investigational drug protocol.
  * Use of any prohibited medications within 14 days or 5 half-lives (whichever is longer) of the baseline visit.
* Parent or legal guardian who, in the opinion of the investigator, is unable or unlikely to comply with the administration schedule and study evaluations or are unable or unwilling to apply the study drug.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Participants with treatment-emergent adverse events (TEAEs) | Screening through 30-37 days after end of treatment, up to approximately 12 weeks.
  A TEAE is any adverse event (AE) either reported for the first time or worsening of a pre-existing event after first application of study drug.

SECONDARY OUTCOMES:
Plasma concentrations of ruxolitinib for Cohorts 1 and 2 | Day 1, Day 15, and Day 29
  Venous blood samples will be collected to assess the PK of ruxolitinib .
Plasma concentrations of ruxolitinib for Cohorts 3, 4, 5 and 6 | Day 1, Day 10, and Day 29
  Venous blood samples will be collected to assess the PK of ruxolitinib .

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kuligowski, MD, PhD, MBA, Study Director — Incyte Corporation
Locations (23):
- United States (23):
  - Cahaba Dermatology, Hoover, Alabama
  - Desert Sky Dermatology, Gilbert, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Orange County Research Center, Anaheim, California
  - Children'S Hospital Los Angeles Specialt, Los Angeles, California
  - Rady Children'S Hospital - San Diego, San Diego, California
  - National Jewish Health, Denver, Colorado
  - Olympian Clinical Research, Largo, Florida
  - Acevedo Clinical Research, Miami, Florida
  - Floridian Research Institute Llc, Miami, Florida
  - Rm Medical Research Inc, Miami, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Iact Health, Columbus, Georgia
  - Advanced Clinical Research, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - The Indiana Clincal Trials Center, Plainfield, Indiana
  - David Fivenson, Md, Pllc, Ann Arbor, Michigan
  - Wake Research Associates Llc, Raleigh, North Carolina
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Cyn3Rgy Research - Clinedge - Ppds, Gresham, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leung DYM, Paller AS, Zaenglein AL, Tom WL, Ong PY, Venturanza ME, Kuligowski ME, Li Q, Gong X, Lee MS. Safety, pharmacokinetics, and efficacy of ruxolitinib cream in children and adolescents with atopic dermatitis. Ann Allergy Asthma Immunol. 2023 Apr;130(4):500-507.e3. doi: 10.1016/j.anai.2022.12.033. Epub 2022 Dec 28. PMID 36586583